CLINICAL TRIAL: NCT00478985
Title: Evaluation of the Persistence of the Complete Molecular Remission After Stopping Imatinib Chronic Myeloid Leukemia (STIM)
Brief Title: Evaluation of the Persistence of the Complete Molecular Remission After Stopping Imatinib Chronic Myeloid Leukemia
Acronym: STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2006/06
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: Leukemia; Adult Chronic; Myeloid
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Imatinib treatment ending
  Interventions: Behavioral: Imatinib ending

INTERVENTIONS:
Behavioral: Imatinib ending — Interruption of the treatment by Imatinib

SUMMARY:
The first purpose of this study is to evaluate the persistence of the complete molecular remission in patients with Chronic Myeloid Leukemia after stopping imatinib treatment (determine by Reverse Transcription real-time Polymerase Chain Reaction (RT-PCR) negative for bcr-abl transcripts). The second purpose is to determine clinicals and biologicals factors associated with the persistent complete molecular remission.

DETAILED DESCRIPTION:
Principal Objective : To evaluate the complete molecular remission persistence after stopping imatinib during six months as measured by RT-PCR negative for bcr-abl transcripts in patients with Chronic Myeloid Leukemia .

Secondary Objective :

* To determine clinicals factors associated with complete molecular remission before and after stopping imatinib in patients with Chronic Myeloid Leukemia.
* To determine the biologics factors (immunologic and molecular) associated with complete molecular remission before and after stopping imatinib in patients with Chronic Myeloid Leukaemia.
* To determine the molecular relapse level after more than six month of persistent complete molecular remission without imatinib.
* To determine the complete molecular remission length.
* To evaluate medical and economical impact of stopping imatinib treatment.

Study design : multicentric trial

ELIGIBILITY:
Inclusion Criteria:

* Patients must have reached their 18th birthday
* Women of childbearing potential must agree to use effective methods of contraception
* Patients must be affiliated to a social security regime
* Patients must have received imatinib therapy for at least 36 months.
* Patients must be in complete molecular remission during at least two consecutive years with at least five RT-PCR negative measures for bcr-abl transcripts.
* Patients must be HIV, HCV and HBV negatives
* Patients who have molecular follow-up realized in accordance with international recommendations
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent.

Exclusion Criteria:

* Patients who are protected by the law. Patients who are unable to give their consent to participate to the study.
* Patients who have pathologies or treatments that are able to enhance the potential relapse risk after stopping imatinib. Patients who have pathologies or treatments which able to interfere with immunologic study (excepted IFN α):

Corticosteroids or other immuno suppressors Other concomitant malign pathology treated by chemotherapy or radiotherapy Previous or programmed Haematopoietic Stem Cell allogreffe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of complete molecular remission persistence as measured by RT-PCR negative for bcr-abl transcripts | Every month during the first year and every two months during the second year

SECONDARY OUTCOMES:
T lymphocytes differenciation and proliferation analyse / cytokines production analyse | first visit, M2,M4,M6,M9,M12,M18,M24
T lymphocytes apoptosis analyse | first visit
Haemogramme analyse | every months during two years
Clinical exam | every three months during the first year and every four months during the second year

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier MAHON, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (24):
- France (24):
  - University Hospital Angers, Angers, Angers
  - Hôpital Morvan, Brest, Brest
  - Hôpital Henri-Mondor, Créteil, Créteil
  - Hôpital Claude Huriez, Lille, Lille
  - University Hospital Hôtel-Dieu, Nantes, Nantes
  - Hôpital Saint Louis, Paris, Paris
  - University Hospital Poitiers, Poitiers, Poitiers
  - University Hospital Toulouse, Purpan, Toulouse, Toulouse
  - University Hospital Brabois, Vandœuvre-lès-Nancy, Vandoeuvre Les Nancy
  - Institut Bergonié, Bordeaux
  - University Hospital Bordeaux, Groupe Hospitalier Pellegrin, Bordeaux
  - CHU de Grenoble, Grenoble
  - Centre hospitalier-service de médecine interne Onco-Hématologique, La Roche-sur-Yon
  - Hôpital André Mignot, Le Chesnay
  - Hôpital Bicêtre, AP-HP, Le Kremlin-Bicêtre
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmet, Marseille
  - CHR de Metz-Thionville, Metz
  - Centre Hospitalier de Nevers, Nevers
  - University Hospital Nice, Nice
  - Hôpital Necker-Enfants Malades, Paris
  - Haut Lévêque Hospital, Pessac
  - University Hospital Strasbourg, Hôpital Civil, Strasbourg
  - Centre Hospitalier Bretagne Atlantique, Vannes

REFERENCES:
- [Derived] Mahon FX, Dulucq S, Rea D, Nicolini FE, Rigal-Huguet F, Machova Polakova K, Dubruille V, Noel MP, Ianotto JC, Villemagne B, Cayssials E, Park S, Rousselot P, Etienne G. Extended long-term follow-up and the survival of Stop Imatinib study. Blood Neoplasia. 2025 Oct 27;3(1):100177. doi: 10.1016/j.bneo.2025.100177. eCollection 2026 Feb. PMID 41574312
- [Derived] Rea D, Henry G, Khaznadar Z, Etienne G, Guilhot F, Nicolini F, Guilhot J, Rousselot P, Huguet F, Legros L, Gardembas M, Dubruille V, Guerci-Bresler A, Charbonnier A, Maloisel F, Ianotto JC, Villemagne B, Mahon FX, Moins-Teisserenc H, Dulphy N, Toubert A. Natural killer-cell counts are associated with molecular relapse-free survival after imatinib discontinuation in chronic myeloid leukemia: the IMMUNOSTIM study. Haematologica. 2017 Aug;102(8):1368-1377. doi: 10.3324/haematol.2017.165001. Epub 2017 May 18. PMID 28522576
- [Derived] Mahon FX, Rea D, Guilhot J, Guilhot F, Huguet F, Nicolini F, Legros L, Charbonnier A, Guerci A, Varet B, Etienne G, Reiffers J, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chroniques. Discontinuation of imatinib in patients with chronic myeloid leukaemia who have maintained complete molecular remission for at least 2 years: the prospective, multicentre Stop Imatinib (STIM) trial. Lancet Oncol. 2010 Nov;11(11):1029-35. doi: 10.1016/S1470-2045(10)70233-3. Epub 2010 Oct 19. PMID 20965785